CLINICAL TRIAL: NCT01415102
Title: A Double Blind (3rd Party Open), Randomised, Placebo-Controlled, Dose Escalation Study To Investigate The Safety, Toleration, And Pharmacokinetics Of Single Inhaled Doses Of Pf-05212372 In Healthy Subjects
Brief Title: A First In Human Study In Healthy People To Evaluate Safety, Toleration And Time Course Of Plasma Concentration Of Single Inhaled Doses Of PF-05212372.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2031001
Record Dates: First submitted 2010-09-29; First posted 2011-08-11 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Phase 1; Single Dose; Safety; Toleration; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects will be assigned to receive either PF-05212372 or placebo in each period
  Interventions: Drug: PF-05212372; Drug: Placebo
- Cohort 2 (Experimental): Subjects will be assigned to receive either PF-05212372 or placebo in each period
  Interventions: Drug: PF-05212372; Drug: Placebo

INTERVENTIONS:
Drug: PF-05212372 — Inhaled. Dose Level 1: 50 ug
  Arms: Cohort 1
Drug: PF-05212372 — Inhaled. Dose Level 2 - Dose to be selected based upon safety/tolerability/PK at preceding dose
  Arms: Cohort 1
Drug: PF-05212372 — Inhaled. Dose Level 3 - Dose to be selected based upon safety/tolerability/PK at preceding dose
  Arms: Cohort 1
Drug: PF-05212372 — Inhaled. Dose Level 4 - Dose to be selected based upon safety/tolerability/PK at preceding dose
  Arms: Cohort 1
Drug: Placebo — Inhaled
  Arms: Cohort 1
Drug: PF-05212372 — Inhaled. Dose Level 5 - Dose to be selected based upon safety/tolerability/PK at preceding dose
  Arms: Cohort 2
Drug: PF-05212372 — Inhaled. Dose Level 6 - Dose to be selected based upon safety/tolerability/PK at preceding dose
  Arms: Cohort 2
Drug: PF-05212372 — Inhaled. Dose Level 7 - Dose to be selected based upon safety/tolerability/PK at preceding dose
  Arms: Cohort 2
Drug: Placebo — Inhaled
  Arms: Cohort 2

SUMMARY:
The purpose of this study in healthy people is to evaluate safety, toleration and time course of plasma concentration of single inhaled doses of PF-05212372.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* Treatment with an investigational drug within the past 30 days (or local regulations) or 5 half-lives preceding the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 14 days
Plasma pharmacokinetics | up to 72 hours post dose
Urine pharmacokinetics | up to 24 hours post dose
Urine Pharmacodynamics | up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2031001&StudyName=A%20First%20In%20Human%20Study%20In%20Healthy%20People%20To%20Evaluate%20Safety%2C%20Toleration%20And%20Time%20Course%20Of%20Plasma%20Concentration%20Of%20Single%20Inhaled%20